CLINICAL TRIAL: NCT00913146
Title: Can Treatment of Malaria be Restricted to Parasitologically Confirmed Malaria? A School-Based Prospective, Exposed/Non Exposed to Fever, Study in Benin.
Brief Title: Can Treatment of Malaria be Restricted to Parasitologically Confirmed Malaria?
Status: Completed | Type: Observational
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: Institut de Médecine et d'Epidémiologie Appliquée - Fondation Internationale Léon M'Ba (Other)
Responsible Party: Jean-François Faucher, MD, Institut de Recherche pour le Developpement
Other Study IDs: IMEA5982FAU90
Record Dates: First submitted 2009-06-03; First posted 2009-06-04 (Estimated); Last update posted 2009-06-04 (Estimated); Status verified 2009-06

CONDITIONS: Malaria
Keywords: Management of fever; Malaria; Malaria rapid diagnostic test; Clinical trial
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood dried on filter papers
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- index: child with fever and a negative malaria RDT
- control: apparently healthy child with a negative RDT

SUMMARY:
The investigators performed a prospective study, in order to assess the feasibility and safety of restricting antimalarials to rapid diagnostic test (RDT)-confirmed cases in children aged 5 to 15 years-old

DETAILED DESCRIPTION:
This study was designed to measure the incidence of malaria attacks during a 2-week follow-up period in 2 populations of patients. First, an index group (IG, exposed to fever) constituted by schoolchildren attending the school nursery for fever and not diagnosed malaria, based on a negative HRP2-based RDT. Second, a control group (CG, not exposed to fever) constituted of apparently healthy schoolchildren paired with index cases on gender, age, week of inclusion and malaria status (ie: negative HRP2-based RDT).

In a pragmatic purpose, the subjects were selected for inclusion if no malaria diagnosis was made by the means accessible to a clinician in routine practice, i.e., RDT and body temperature assessment. During the follow-up, malaria was defined as the association of fever and parasitemia, using any malaria diagnostic method, whatever its availability on the field: (blood smear and/or PCR).

Hence, the primary objective of the study was to show that applying the algorithm of management of fevers in the school setting is safe, in the way it does not lead to an excessive number of undiagnosed (and thus untreated) malaria attacks, by comparing the number of malaria attacks between the two groups (exposed and non exposed to fever).

The secondary objective was to compare malaria incidence between children at high risk for malaria during follow-up in the IG and CG respectively. Children at high risk for malaria in these 2 groups were defined by the detection of Plasmodium falciparum infection at enrollment, using the most sensitive diagnostic tool currently available (i.e., PCR). Based on data from the literature, we estimated to about 15% the proportion of children attending for fever with a negative RDT and a positive PCR for malaria, and we assumed this proportion to be roughly the same in apparently healthy children. Twenty-eight children at high risk for malaria in each group (corresponding to187 children in each group) are needed to detect an 8% difference in proportion between the 2 groups (α = 0.05 and β = 0.8). Assuming a maximum of 5% in the dropout rate, we aimed at including a minimum of 200 children in each group.

Study site: This study was performed from February through June 2008 in 4 schools, located at Allada, Southern-Benin, where malaria transmission is intense and perennial. Altogether, the 4 study schools received about 2600 schoolchildren of 5 years-old and above.

Conduct of the study: Ethical clearance was obtained from the Faculty of Medicine ethics committee, Benin National University, Cotonou. Children attended school nurseries on their own, or led by their parents/guardians. Care was provided for any child from a school participating to the study. Children from the IG were included and actively followed only if individual informed consent was obtained (within 24 hours from the initial visit) from a parent or guardian. Asymptomatic children were screened for the CG on gender, age, week of inclusion. The first child with a negative RDT and for whom an informed consent was obtained, was included in the CG. Asymptomatic children (screened for inclusion into the CG) and with a positive RDT were advised to quickly attend at the school nursery as soon as symptoms of malaria would appear. Children treated for malaria within the prior month were not included in either group.

All children were examined by a study nurse. Children with danger signs were referred to a health centre. Children attending the school nurseries were managed for fever only if fever was stated (tympanic temperature at 37.8°C or above) or if an history of fever in the preceding 24 hours was reported. For each schoolchild managed for fever, a RDT (Paracheck®, ORCHID Diagnostics) was performed and children were given artemether-lumefantrine (AL) if the RDT result was positive, according to national guidelines in this age group. At enrolment and during follow-up, medications with antimalarial activity for the treatment of non malarial illnesses were avoided when acceptable alternatives were available.

Follow-up visits were on day 3, 7 and 14. A blood smear and a blood spot were collected at enrolment and at each scheduled visit. An additional blood spot for pharmacological data was collected for 100 children in each group on day 0 and day 14. When fever was reported and/or stated at a follow-up visit, a RDT was performed.

We estimated the number of undiagnosed P falciparum malaria at enrolment, by taking into account both baseline data (all cases with P falciparum parasitemia >1000/µL) and follow-up data with fever with concomitant occurrence of at least one test (including PCR) positive for a P falciparum infection.

Laboratory analysis: RDTs were red by the study nurse, as recommended by manufacturer 15 minutes after it was performed. Microscopy examination was done retrospectively (patients were managed according to RDT results in terms of antimalarials prescriptions and IG or CG group assignment) and blinded to the patient's identity.

DNA was prepared from blood collected at day 0 and on the last day of follow-up, as well as at occurrence of fever during follow-up.

On day 0 and day 14 in the 100 first children from each group, whole blood was sampled on filter paper spots and dried at room temperature. Using these dried blood spot (DBS), chloroquine (and monodesethylchloroquine) and quinine were detected by high pressure liquid chromatography with UV detection to 254 nm using ammonium acetate (40 mM, pH =5.5)/acetonitrile (85/15 % v/v).

Statistics: Parametric tests (Pearson's chi-square and chi-square for the comparison of crude rates) and non-parametric (Fischer) tests were used. A logistic regression on PCR positivity at enrollment was performed, taking into account variables likely to influence the malarial status: gender, age, school, clinical status, declared bednet use.

ELIGIBILITY:
Inclusion Criteria in the index group:

* School children aged 5 to 15 years.
* Tympanic temperature at 37.8°C or above, or if a history of fever in the preceding 24 hours was reported.
* A negative malaria (Paracheck® Plasmodium falciparum) RDT.
* Informed consent.
* Asymptomatic children were screened for the Control Group on gender, age, week of inclusion. The first child with a negative RDT and for whom an informed consent was obtained, was included in the CG.

Exclusion Criteria:

* Adequate malaria treatment within a month prior screening.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 2600 schoolchildren of 5 years-old and above
Sampling Method: Non-Probability Sample
Enrollment: 484 (Actual)
Dates: Start 2008-02; Primary Completion 2008-06 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
malaria incidence in the 2 groups (index and control) | after 14 days of follow-up

SECONDARY OUTCOMES:
malaria incidence in children with a positive Plasmodium falciparum PCR at baseline | after 14 days of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Faucher, MD, PhD, Principal Investigator — IRD
Locations (1):
- Centre de Santé de Commune, Allada, Benin

REFERENCES:
- [Background] Njama-Meya D, Clark TD, Nzarubara B, Staedke S, Kamya MR, Dorsey G. Treatment of malaria restricted to laboratory-confirmed cases: a prospective cohort study in Ugandan children. Malar J. 2007 Jan 21;6:7. doi: 10.1186/1475-2875-6-7. PMID 17239256
- [Background] Msellem MI, Martensson A, Rotllant G, Bhattarai A, Stromberg J, Kahigwa E, Garcia M, Petzold M, Olumese P, Ali A, Bjorkman A. Influence of rapid malaria diagnostic tests on treatment and health outcome in fever patients, Zanzibar: a crossover validation study. PLoS Med. 2009 Apr 28;6(4):e1000070. doi: 10.1371/journal.pmed.1000070. Epub 2009 Apr 28. PMID 19399156